CLINICAL TRIAL: NCT00300378
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of 2 Fixed Doses (50 mg, 100 mg) of Desvenlafaxine Sustained-Release Tablets in Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating the Efficacy and Safety of Desvenlafaxine Tablets in Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A1-333
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Adult; Outpatients
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Desvenlafaxine Succinate

INTERVENTIONS:
Drug: desvenlafaxine 50 mg
Drug: desvenlafaxine 100 mg

SUMMARY:
The primary objective is to compare the antidepressant efficacy, safety, and tolerability of DVS SR versus placebo in subjects with Major Depressive Disorder. Additional objectives include testing both general and functional quality-of-life outcomes and satisfaction with therapy reported by the subject.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of MDD
* Depressive symptoms for at least 30 days before the screening visit.

Exclusion Criteria:

* Treatment with DVS SR at any time in the past.
* Known hypersensitivity to venlafaxine
* Significant risk of suicide based on clinical judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2006-03; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the change from baseline on the 17-item of the Hamilton Depression rating scale (HAM-D17 score) at the final on therapy evaluation

SECONDARY OUTCOMES:
The Global Clinical Improvement will be the key secondary efficacy variable.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Estonia, Latvia, Lithuania, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Romania, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Finland, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Croatia, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Slovakia, DIS-WP-BV-EUBV01-Medical@wyeth.com
Locations (39):
- Croatia (3):
  - Rijeka
  - Split
  - Zagreb
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (8):
  - Espoo
  - Helsinki
  - Joensuu
  - Kuopio
  - Oulu
  - Rauma
  - Salo
  - Turku
- France (7):
  - Caen
  - Dole
  - Douai
  - Mulhouse
  - Orvault
  - Rennes
  - Tours
- Latvia (4):
  - Jelgava
  - Liepāja
  - Riga
  - Strenči
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (3):
  - Lubiąż
  - Tuszyn
  - Żuromin
- Romania (2):
  - Bucharest
  - Craiova
- Slovakia (3):
  - Bojnice
  - Bratislava
  - Rimavská Sobota
- South Africa (4):
  - Bloemfontein
  - Cape Town
  - Durban
  - Pretoria

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] Soares CN, Zhang M, Boucher M. Categorical improvement in functional impairment in depressed patients treated with desvenlafaxine. CNS Spectr. 2019 Jun;24(3):322-332. doi: 10.1017/S1092852917000633. Epub 2017 Nov 15. PMID 29140227
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Soares CN, Endicott J, Boucher M, Fayyad RS, Guico-Pabia CJ. Predictors of functional response and remission with desvenlafaxine 50 mg/d in patients with major depressive disorder. CNS Spectr. 2014 Dec;19(6):519-27. doi: 10.1017/S1092852914000066. Epub 2014 Feb 26. PMID 24571916